CLINICAL TRIAL: NCT01436227
Title: A Phase II Trial of Pazopanib in Von Hippel-Lindau Syndrome
Brief Title: Pazopanib Hydrochloride in Treating Patients With Von Hippel-Lindau Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0465; NCI-2011-03285 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0465 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Von Hippel-Lindau Syndrome
MeSH Terms: conditions — von Hippel-Lindau Disease | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28. Treatment repeats every 4 weeks for up to 24 weeks in the absence of disease progression or unacceptable toxicity. Patients benefitting from treatment may continue pazopanib hydrochloride in the absence of disease progression.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient

SUMMARY:
This phase II trial studies the side effects and how well pazopanib hydrochloride works in treating patients with von Hippel-Lindau syndrome. Pazopanib hydrochloride may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate safety and efficacy of treatment with pazopanib hydrochloride (pazopanib) for 6 months in patients with von Hippel-Lindau syndrome (VHL) who have a measurable VHL related lesion.

SECONDARY OBJECTIVES:

I. Evaluate rate of growth over time in target lesions before and after pazopanib treatment.

II. Evaluate need for surgical intervention over time in patients who receive pazopanib and compare to rate prior to receipt of drug.

III. Create an annotated tissue resource from patients with VHL for use in future research related to cancer.

PRECLINICAL OBJECTIVES:

I. Evaluate circulating factors in patients with VHL undergoing treatment with pazopanib.

II. Evaluate relationship between VHL genotype and response to pazopanib.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Treatment repeats every 4 weeks for up to 24 weeks in the absence of disease progression or unacceptable toxicity. Patients benefitting from treatment may continue pazopanib hydrochloride in the absence of disease progression.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up; procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Genetically confirmed diagnosis of VHL or measurable disease consistent with the clinical diagnosis of VHL
* At least one measurable VHL related lesion, which is undergoing surveillance, and patient is not at immediate risk of needing intervention for this or other lesions; biopsy is not required given the known likely etiology and natural history in the setting of a positive genetic test

  * Brain: asymptomatic hemangioblastoma, >= 0.5 cm
  * Spine: asymptomatic hemangioblastoma, >= 0.5 cm
  * Renal: solid mass suspicious for renal cell carcinoma (RCC) >= 1 cm or cystic mass (Bosniak 3-4) >= 1 cm
  * Pancreas: solid mass >= 1 cm and =< 3 cm suspicious for neuroendocrine tumor, or neuroendocrine tumor > 3 cm but not considered operable
  * Eye: asymptomatic peripapillary and/or macular hemangioblastoma, any size
  * Adrenal: asymptomatic or controlled pheochromocytoma greater than 1 cm in size
* Patients may have received prior VHL-related systemic therapy, provided not within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Hemoglobin >= 9 g/dL (5.6 mmol/L)

  * Subjects may not have had a transfusion within 7 days of screening assessment
* Platelets >= 100 X 10^9/L
* Prothrombin time (PT) or international normalized ratio (INR) =< 1.2 X upper limit of normal (ULN)

  * Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation or if they are on low molecular weight heparin
* Activated partial thromboplastin time (aPTT) =< 1.2 X ULN
* Total bilirubin =< 1.5 X ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.0 X ULN

  * Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted
* Serum creatinine =< 2.0 mg/dL (133 umol/L) OR, if > 2.0 mg/dL: calculated creatinine clearance (ClCR) >= 50 mL/min
* Urine protein to creatinine ratio (UPC) < 1

  * If UPC >= 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value < 1 g to be eligible
* A female is eligible to enter and participate in this study if she is of: non-childbearing potential including

  * Any female who has had a surgical procedure rendering her incapable of becoming pregnant
  * Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40 pg/mL (< 140 pmol/L)
  * Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT; childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception GlaxoSmithKline (GSK) acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
    * Oral contraceptive
    * Injectable progestogen
    * Implants of levonorgestrel
    * Estrogenic vaginal ring
    * Percutaneous contraceptive patches
    * Intrauterine device (IUD)
    * Male partner sterilization
    * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository); female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug

Exclusion Criteria:

* Prior malignancy. Subjects who have had another non VHL related malignancy and have been disease-free for 2 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel
* Presence of uncontrolled infection
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension (defined as systolic blood pressure [SBP] of >= 140 mmHg or diastolic blood pressure [DBP] of >= 90 mmHg); Note: initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry; blood pressure (BP) must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP/DBP values from each BP assessment must be < 140/90 mmHg in order for a subject to be eligible for the study
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months; Note: subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
* Evidence of active bleeding or bleeding diathesis
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Unable or unwilling to discontinue use of prohibited medications list for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
* Treatment with any of the following anti-cancer therapies:

  * Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
  * Chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
* Any ongoing toxicity from prior investigational therapy that is > grade 1 and/or that is progressing in severity, except alopecia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jonasch E, McCutcheon IE, Gombos DS, Ahrar K, Perrier ND, Liu D, Robichaux CC, Villarreal MF, Weldon JA, Woodson AH, Pilie PG, Fuller GN, Waguespack SG, Matin SF. Pazopanib in patients with von Hippel-Lindau disease: a single-arm, single-centre, phase 2 trial. Lancet Oncol. 2018 Oct;19(10):1351-1359. doi: 10.1016/S1470-2045(18)30487-X. Epub 2018 Sep 17. PMID 30236511
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2012 to August 2016, patients were recruited from the outpatient clinics for Genitourinary Medical Oncology at MD Anderson Cancer Center in Houston, Texas who have been diagnosed with Von Hippel-Lindau Syndrome.
Pre-assignment Details: 32 subject enrolled
Groups:
- Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28: Pazopanib 800mg PO Daily
Period: Overall Study
Arm/Group | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28
Started | 32
Completed | 6
Not Completed | 26
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 7
Not completed — Disease progression, relapse | 6

BASELINE CHARACTERISTICS:
Population: All dosed participants
Arm/Group | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response + Partial Response)
Description: Overall response rate (complete response + partial response) Determined by the Response Evaluation Criteria in Solid Tumors. Estimated with its corresponding 95% posterior credible interval.
Time Frame: At 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28
Number analyzed (Participants) | 31
Participants | 13

2. Primary Outcome: Progressive Disease Rate
Description: Progressive disease rate
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28
Number analyzed (Participants) | 31
Participants | 6

3. Primary Outcome: Drug Discontinuation Due to Toxicity
Description: Drug discontinuation due to toxicity
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28
Number analyzed (Participants) | 31
Participants | 7

4. Primary Outcome: Time to Progression (TTP)
Description: TTP will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between prognostic groups. Regression analyses of survival data based on the Cox proportional hazards model will be conducted on TTP. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure that the models are appropriate.
Time Frame: Up to 24 weeks
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28
Number analyzed (Participants) | 32
Days | NA (NA) — There is no data to report due to median PFS not being reached.

ADVERSE EVENTS:
Time Frame: From first dose until 30 days after last dose of drug, up to 28 weeks.
Description: Death or life-threatening events that place the patient at immediate risk of death (excluding those that could lead to death in a more severe form). Includes inpatient hospitalization, extended hospitalization, significant incapacity, or major disruption of normal life functions. Also includes congenital anomalies or birth defects.
Arm/Group | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28
All-Cause Mortality (participants affected / at risk) | 1/32
Serious Adverse Events (participants affected / at risk) | 12/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28 (N=32)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Appendicitis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Blood and lymphatic system disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, Fatigue weakness (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 2
Nervous system disorders - Other, increased right hand weakness and difficulty performing ADL. (Nervous system disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Stroke (Nervous system disorders) | 1
Surgical and medical procedures - Other, stereotactic radiosurgery (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pazopanib Hydrochloride) Patients Receive Pazopanib Hydrochloride PO QD on Days 1-28 (N=32)
Abdominal pain (Gastrointestinal disorders) | 4
Activated partial thromboplastin time prolonged (Investigations) | 2
Akathisia (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 19
Alkaline phosphatase increased (Investigations) | 6
Allergic reaction (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9
Anemia (Blood and lymphatic system disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 5
Anxiety (Psychiatric disorders) | 4
Appendicitis (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 19
Ataxia (Nervous system disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bloating (Gastrointestinal disorders) | 1
Blood bilirubin increased (Blood and lymphatic system disorders) | 7
Blurred vision (Eye disorders) | 6
Cholesterol high (Investigations) | 2
Colitis (Gastrointestinal disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 9
Depression (Psychiatric disorders) | 11
Diarrhea (Gastrointestinal disorders) | 26
Dizziness (Nervous system disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema limbs (General disorders) | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Eye disorders - Other, specify (Eye disorders) | 2
Facial nerve disorder (General disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 27
Fever (General disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flashing lights (Eye disorders) | 1
Floaters (Eye disorders) | 2
Flu like symptoms (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gait disturbance (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
General disorders and administration site conditions - Other, specify (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
GGT increased (Investigations) | 2
Glucose intolerance (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 14
Hearing impaired (Ear and labyrinth disorders) | 4
Hematuria (Renal and urinary disorders) | 1
Hemoglobinuria (Renal and urinary disorders) | 2
Hot flashes (Vascular disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 23
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 17
Hyperthyroidism (Endocrine disorders) | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypothyroidism (Endocrine disorders) | 1
Immune system disorders - Other, specify (General disorders) | 1
Insomnia (Psychiatric disorders) | 6
Intracranial hemorrhage (Nervous system disorders) | 1
Investigations - Other, specify (General disorders) | 3
Irregular menstruation (General disorders) | 2
Libido decreased (General disorders) | 1
Lipase increased (Investigations) | 4
Localized edema (General disorders) | 1
Lymphocyte count decreased (Investigations) | 3
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 10
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 18
Neck pain (Musculoskeletal and connective tissue disorders) | 8
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 8
Nystagmus (Nervous system disorders) | 2
Optic nerve disorder (Eye disorders) | 3
Pain (General disorders) | 6
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Penile infection (Infections and infestations) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8
Personality change (Nervous system disorders) | 1
Photophobia (Eye disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 7
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 2
Serum amylase increased (Investigations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 16
Somnolence (Nervous system disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Suicidal ideation (Nervous system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 6
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 2
Urinary urgency (Renal and urinary disorders) | 1
Vaginal infection (Renal and urinary disorders) | 1
Vaginal inflammation (Renal and urinary disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Watering eyes (Eye disorders) | 1
Weight loss (General disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Investigations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT01436227/Prot_SAP_000.pdf